CLINICAL TRIAL: NCT06043336
Title: A Comparative Study Between Palonosetron vs the Combination of Granisetron and Dexamethasone in Preventing Postoperative Nausea and Vomiting in Laparoscopic Cholecystectomy.
Brief Title: Palonosetron vs Combination of Granisetron and Dexamethasone in Preventing PONV in Laparoscopic Cholecystectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FF-2018-209; Fundamental data (Other: Faculty of Medicine, Universiti Kebangsaan Malaysia)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Granisetron; Palonosetron

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group B (Active Comparator): Group B received intravenous (IV) dexamethasone 4 mg after intubation & IV granisetron 1 mg at the end of surgery
  Interventions: Drug: Dexamethasone, granisetron & palonosetron
- Group A (Experimental): Group A received 1 ml of intravenous (IV) 0.9% saline after intubation and IV palonosetron 0.075 mg at the end of operation.
  Interventions: Drug: Dexamethasone, granisetron & palonosetron

INTERVENTIONS:
Drug: Dexamethasone, granisetron & palonosetron — . Group A received 1 ml of intravenous (IV) 0.9% saline after intubation and IV palonosetron 0.075 mg at the end of operation. Group B received IV dexamethasone 4 mg after intubation and IV granisetron 1 mg at the end of surgery

SUMMARY:
This is a prospective, randomized, double-blinded study comparing the post-operative nausea vomiting (PONV) profile following administration of intraoperative palonosetron alone and the combination of granisetron and dexamethasone in moderate to high-risk patients undergoing elective laparoscopic cholecystectomy.

Patients aged 18-65 years with American Society of Anesthesiologists physical status I or II were randomized into two groups. Group A received 1 ml of intravenous (IV) 0.9% saline after intubation and IV palonosetron 0.075 mg at the end of operation. Group B received IV dexamethasone 4 mg after intubation and IV granisetron 1 mg at the end of surgery. The occurrence of PONV and the need for rescue antiemetics were assessed at 30 minutes, 4, 24 and 48 hours post-anesthesia. A complete response towards the study drugs was considered when patients did not experience PONV and did not require rescue antiemetics. The side effects of the study drugs were evaluated. Patient satisfaction with the anti-emetics administered was assessed.

These parameters were compared between Group A and Group B: the occurrence of PONV, the need of rescue antiemetics, the side effects of the study drugs and patient satisfaction with the anti-emetics administered.

DETAILED DESCRIPTION:
This prospective double-blinded, randomized controlled study was conducted at Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia, Malaysia after obtaining approval from the Institutional Ethics Committee of Universiti Kebangsaan Malaysia (UKM).

Patients aged 18 to 65 years old, American Society of Anesthesiologists (ASA) physical status I or II, scheduled for elective laparoscopic cholecystectomy under general anesthesia were recruited using convenient sampling. Patients with heart diseases, prolonged QT syndrome, a family history of sudden death, known allergies, or contraindications to the study drugs were excluded. No premedication was administered to the patients, and an intravenous (IV) drip was not started preoperatively.

After obtaining written informed consent, patients were randomized to one of two groups using computer-generated random numbers. Group A received IV palonosetron 0.075 mg, and Group B received IV granisetron 1 mg and IV dexamethasone 4 mg as antiemetics.

Patients were fasted for at least 6 hours prior to surgery. In the operating room, standard monitoring was applied to every patient, including continuous electrocardiography (ECG), non-invasive blood pressure monitoring (NIBP), pulse oximetry, capnography with multi-gas analyzer including minimum alveolar concentration (MAC), and monitoring of all gas levels.

Patients were pre-oxygenated with oxygen. Induction of anesthesia was conducted using IV fentanyl 2 mcg/kg and IV propofol 2 mg/kg. Upon loss of consciousness, IV rocuronium 0.6 mg/kg was administered to facilitate endotracheal intubation, following which patients were mechanically ventilated with a mixture of oxygen and air. Anesthesia was maintained with sevoflurane at MAC of 1.0 to 1.2. Ventilation parameters were adjusted to maintain normocapnia (end-tidal carbon dioxide of 35-40 mmHg) and saturation of oxygen above 96%.

Group A patients received 1 ml of IV 0.9% saline while Group B patients received IV dexamethasone 4 mg after intubation. The amount of IV morphine given to the patients intraoperatively was recorded and did not exceed 0.1 mg/kg. Rescue analgesia with IV fentanyl was administered if needed, not exceeding 100 mcg. The surgeon infiltrated 10 ml of levobupivacaine 0.5% into the incisions at the end of surgery. Patients were kept adequately hydrated throughout the surgery with an IV drip of 2 ml/kg/h as maintenance, any fluid deficit was replaced. Pneumoperitoneum in laparoscopic procedure was achieved by carbon dioxide insufflation with intra-abdominal pressure of less than 14 mmHg.

Thirty minutes prior to the end of the surgery, Group A received a slow bolus of IV palonosetron 0.075 mg, while Group B received a slow bolus of IV granisetron 1 mg. Intravenous neostigmine 0.05 mg/kg and IV atropine 0.02 mg/kg were administered as a reversal agent. The pneumoperitoneum was evacuated by the surgeon, and the nasogastric tube was suctioned and removed before extubation. The patients were transferred to the recovery bay after extubation. Rescue analgesia with IV fentanyl was administered in the recovery bay if needed, not exceeding 50 mcg.

Patients were monitored by blinded anesthetists for nausea and vomiting in four time periods: 30 minutes, 4 hours, 24 hours, and 48 hours post-anesthesia. Nausea was defined as an unpleasant sensation associated with the urge to vomit and its severity was rated by patients on a scale of 0 (no nausea) to 10 (worst possible nausea). Vomiting was defined as the forceful expulsion of gastric contents from the mouth, and the frequency of vomiting was recorded. If a patient experienced severe nausea (nausea score of 4 and more) and vomiting, rescue antiemetic of IV metoclopramide 10 mg was administered. Regular IV metoclopramide was administered if the patient experienced a second episode of vomiting or more. A complete response (free from emesis) was defined as no nausea, no vomiting and no need for any rescue medication. Side effects of the study drugs (palonosetron, granisetron, and dexamethasone) such as headache, constipation, dizziness, bloatedness, and palpitation were recorded. At the end of the study, patients were asked if they were satisfied with the antiemetics given to them. Patient satisfaction was assessed by using a Likert scale, which included a five-point scale; very satisfied, satisfied, neutral, dissatisfied, and very dissatisfied. Surgeries that lasted more than four hours, required conversion to open cholecystectomy or other procedures, and severe PONV that did not resolve with rescue anti-emetics were considered dropouts in this study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I or II
* scheduled for elective laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* patients with heart diseases
* patients with prolonged QT syndrome
* patients with a family history of sudden death
* patients with known allergies to dexamethasone, granisetron & palonosetron
* patients with contraindications to dexamethasone, granisetron & palonosetron

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Complete response towards the study drugs | 1 year
  Number of patients who did not experience postoperative vomiting, did not experience postoperative nausea & did not require rescue antiemetics.

SECONDARY OUTCOMES:
The side effects of the study drugs | 1 year
  Number of patients who developed side effects after receiving the study drugs

OTHER OUTCOMES:
Patient satisfaction with the anti-emetics administered | 1 year
  Number of patients who satisfied with the anti-emetics administered

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Budiman, M.D., Principal Investigator — Faculty of Medicine, Universiti Kebangsaan Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No